CLINICAL TRIAL: NCT01828203
Title: Phase III Study of Minocycline in Acute Spinal Cord Injury
Brief Title: Minocycline in Acute Spinal Cord Injury (MASC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rick Hansen Institute (Other)
Collaborators: University of Calgary (Other); Alberta Paraplegic foundation (Unknown)
Responsible Party: Principal Investigator, Steve Casha, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHI-1005
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Spinal Cord Injuries
Keywords: minocycline; randomized control trial; phase 3; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): Minocycline twice daily infused over 30 minutes through central venous access as follows 800 mg + 700 mg on Day 1, 600 mg + 500 mg on Day 2, and 400 mg thereafter from Day 3 thru Day 7
  Interventions: Drug: Minocycline; Procedure: Surgical spinal cord decompression; Procedure: Maintenance of minimum mean arterial pressure (MAP)
- Placebo (Placebo Comparator): 250 ml normal saline and infused over 30 minutes through central venous access twice daily for 7 days
  Interventions: Drug: Placebo; Procedure: Surgical spinal cord decompression; Procedure: Maintenance of minimum mean arterial pressure (MAP)

INTERVENTIONS:
Drug: Minocycline
  Arms: Minocycline
Drug: Placebo
  Arms: Placebo
Procedure: Surgical spinal cord decompression — Surgical decompression by means at the discretion of the clinical management team will occur within 24 hours of injury in all subjects. Stabilization will occur at that time but may also include further interventions at a later time.
Procedure: Maintenance of minimum mean arterial pressure (MAP) — Standardized hemodynamic management protocol aimed at maintaining MAP ≥ 85 mm Hg for 7 days using volume augmentation with isotonic crystalloid followed by inotropic support if needed will be applied to all subjects.

SUMMARY:
The objective of this study is to assess the efficacy of IV minocycline in improving neurological and functional outcome after acute non-penetrating traumatic spinal cord injury (SCI).

The primary hypothesis is that intravenous minocycline twice daily (800 mg initial dose tapered to 400 mg by 100 mg at each dose then administered to the end of day 7) administered to subjects with acute traumatic non-penetrating cervical SCI starting within 12 hours of injury will improve motor recovery as assessed by the International Standards for Neurologic Classification of Spinal Cord Injury - ISNCSCI (a.k.a. ASIA) neurological examination measured between 3 months and 1 year post-injury, compared to placebo.

The secondary hypotheses are that the above minocycline treatment will also results in improvement in ASIA sensory improvement, in ASIA grade and in functional outcome as assessed by Spinal Cord Independence Measure (SCIM) and Short Form 36 (SF-36), compared to placebo. In addition the effect of minocycline on neurological and functional outcome after SCI is expected to be more pronounced in those subjects with motor incomplete SCI compared to those with motor compete SCI. A subgroup analysis will be undertaken to examine this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or over
* Acute traumatic non-penetrating cervical SCI involving neurological levels as defined by the ASIA neurological examination between C0 and C8 and resulting in a detectable change in the ASIA motor assessment
* Patient English speaking and able to provide informed consent
* Randomization and administration of first dose (drug or placebo) within 12 hours of injury.

Exclusion Criteria:

* History of systemic lupus erythematosus (SLE)
* Pre-existing hepatic or renal disease
* Tetracycline hypersensitivity
* Pregnancy or breast feeding
* Isolated radicular motor deficit
* Significant leucopenia (white blood cell count < 1⁄2 times the lower limit of normal) at screening
* Elevated liver function tests (AST, ALT, alkaline phosphatase, or total bilirubin > 2 times the upper limit of normal) at screening
* Presence of systemic disease that might interfere with patient safety, compliance or evaluation of the condition under study (e.g. insulin-dependent diabetes, Lyme disease, clinically significant cardiac disease, HIV, HTLV-1)
* Associated traumatic conditions interfering with informed consent or outcome assessment (e.g. closed head injury, liver contusion)
* Known uncorrected severe coronary artery disease or evidence of active coronary ischemia (ECG changes, positive Troponin) will be excluded, as they may not tolerate the standardized protocol for hemodynamic management

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
ASIA Motor Recovery | assessed at time points: day 1,3,7, week 3,6, month 3,6,12
  Motor recovery (improvement from baseline examination) as assessed by the International Standards for Neurologic Classification of Spinal Cord Injury - ISNCSCI (a.k.a. ASIA) neurological examination measured between 3 months and 1 year post-injury, compared to placebo.

SECONDARY OUTCOMES:
ASIA sensory recovery | assessed at time points: day 1,3,7 week 3,6, months 3,6,12
  Sensory recovery (improvement from baseline) as assessed by the International Standards for Neurologic Classification of Spinal Cord Injury - ISNCSCI (a.k.a. ASIA) neurological examination measured between 3 months and 1 year post-injury, compared to placebo
Spinal cord Independence measure (SCIM) | assessed at time points: week 6, month 3,6,12
  Functional outcome as assessed by the Spinal cord independence Measure assessment at specified time points.
Short Form 36 (SF-36) | assessed at time points: week 6, month 3,6,12
  functional outcome as assessed by the short form 36 (SF-36) quality of Life assessment at specified time points.
ASIA impairment grade | assessed at time points: day 1,3,7 week 3,6 month 3,6,12
  change in ASIA impairment grade at specified time points

OTHER OUTCOMES:
effect of injury severity | as per primary and secondary outcomes
  the sub groups of motor complete (ASIA A and B) and motor incomplete (ASIA C and D) will be examines for each of the primary and secondary outcomes in order to examine the relative efficacy of minocycline in these groups

CONTACTS AND LOCATIONS:
Overall Officials: Steve Casha, MD PhD FRCSC, Principal Investigator — University of Calgary
Locations (7):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta & Royal Alexandra Hospitals, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Hôpital Du Sacré-Cœur de Montréal, Montreal, Quebec

REFERENCES:
- [Background] Casha S, Zygun D, McGowan MD, Bains I, Yong VW, Hurlbert RJ. Results of a phase II placebo-controlled randomized trial of minocycline in acute spinal cord injury. Brain. 2012 Apr;135(Pt 4):1224-36. doi: 10.1093/brain/aws072. PMID 22505632